CLINICAL TRIAL: NCT02580240
Title: Early Initiation of Low-dose Hydrocortisone Treatment for Septic Shock in Adults: a Randomized Clinical Trial
Brief Title: Initiation of Hydrocortisone for the Treatment of Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Qing-quan Lv, Ms Lv, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015KY-127
Record Dates: First submitted 2015-10-18; First posted 2015-10-20 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-04

CONDITIONS: Septic Shock
Keywords: septic shock; hydrocortisone; mortality
MeSH Terms: conditions — Shock, Septic | interventions — Hydrocortisone; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Vials containing normal saline as placebo were identical to those containing hydrocortisone. Placebo administration procedures were similar.
  Interventions: Drug: saline
- hydrocortisone (Experimental): Hydrocortisone was administered 200 mg/d as a continuous infusion for 6d, then tapered off. Once all vasopressors were discontinued, the taper protocol was initiated (half dose for three days, then quarter dose for three days and then stopped).
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone was administered 200 mg/d as a continuous infusion for 6d, then tapered off. Once all vasopressors were discontinued, the taper protocol was initiated (half dose for three days, then quarter dose for three days and then stopped).
  Other Names: cortisol
  Arms: hydrocortisone
Drug: saline — Vials containing normal saline as placebo were identical to those containing hydrocortisone. Placebo administration procedures were similar.
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study : 1）to determine whether hydrocortisone is effective in the treatment of septic shock and 2) to identify the role of timing of low dose hydrocortisone administration in septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years old or older;
2. onset of septic shock within 6 h

Exclusion Criteria:

1. Systemic corticosteroid therapy within the last 3 months before septic shock;
2. high-dose steroid therapy;
3. immunosuppression;
4. refusal of the attending staff or patient family.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qingquan Lv, Master, Principal Investigator — Department of Critical Care Medicine, Northern Jiangsu Province people's hospital
Locations (1):
- Northern Jiangsu Province people's hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lv QQ, Gu XH, Chen QH, Yu JQ, Zheng RQ. Early initiation of low-dose hydrocortisone treatment for septic shock in adults: A randomized clinical trial. Am J Emerg Med. 2017 Dec;35(12):1810-1814. doi: 10.1016/j.ajem.2017.06.004. Epub 2017 Jun 5. PMID 28615145

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Hydrocortisone
Started | 62 | 58
Completed | 60 | 58
Not Completed | 2 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Hydrocortisone | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (16.7) | 68.8 (12.6) | 66.77 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 48
  Male | 37 | 33 | 70
Region of Enrollment [Number; unit: participants]
  China | 60 | 58 | 118

OUTCOME MEASURES:

1. Primary Outcome: 28-day Mortality
Description: Death from any cause at 28 days after the onset of septic shock
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Hydrocortisone
Number analyzed (Participants) | 60 | 58
Participants | 19 | 23

2. Secondary Outcome: All Cause Mortality
Description: Death from any cause at 90 days after the onset of septic shock
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Hydrocortisone
Number analyzed (Participants) | 60 | 58
Participants | 19 | 23

ADVERSE EVENTS:
Time Frame: Adverse Events were classified by onset time （within 60 days after the onset of septic shock）.The adverse events were assessed from date of randomization until 60 days after the onset of septic shock or date of death from any cause, whichever came first, assessed up to 60 days.
Arm/Group | Placebo | Hydrocortisone
All-Cause Mortality (participants affected / at risk) | 19/60 | 23/58
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/58
Other Adverse Events (participants affected / at risk) | 2/60 | 1/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | Hydrocortisone (N=58)
hyperglycemia (Endocrine disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=60) | Hydrocortisone (N=58)
muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No